Document: TDOC-0055319 Version: 1.0; CURRENT; Most-Recent; Effective

Status: Effective

#### **Short Title:**

Effective Date: 25-May-2018

# Statistical Analysis Plan CLL949-C005 / NCT03614130

#### **Full Title:**

# Statistical Analysis Plan CLL949-C005

Protocol Title: Clinical Performance of a Silicone Hydrogel Following Six

Nights of Extended Wear

Project Number:

Protocol TDOC Number: TDOC-0054559

Author:

Template Version:

**Approvals:** See last page for electronic approvals.

Job Notes:

This is the second revision (Version 3.0) of the Statistical Analysis Plan for this study.

Alcon - Business Use Only Statistical Analysis Plan
Document: TDOC-0055319
Status: Effective

Executive Summary:

Key Objectives:

The primary objective is to assess

of the
soft contact lens when worn in an extended wear modality (ie, up to 6 nights of continuous wear) as compared to Biofinity® soft contact lens.

## ${\bf Alcon - Business \ Use \ Only \ \ } {\bf Statistical \ Analysis \ Plan}$


Status: Effective

# **Table of Contents**

Effective Date: 25-May-2018

| Statistic | cal Analysis Plan CLL949-C005 | 1 |
|-----------|-----------------------------------------------------|----|
| Table o | f Contents | 3 |
| List of | Tables | 4 |
| 1 | Study Objectives and Design | 5 |
| 1.1 | Study Objectives | 5 |
| 1.2 | Study Description | |
| 1.3 | Randomization | 5 |
| 1.4 | Masking | 6 |
| 1.5 | Interim Analysis | 6 |
| 2 | Analysis Sets | 6 |
| 2.1 | Safety Analysis Set | 6 |
| 3 | Subject Characteristics and Study Conduct Summaries | 6 |
| 4 | Effectiveness Analysis Strategy | 7 |
| 4.1 | Effectiveness Endpoints | 7 |
| 4.2 | Effectiveness Hypotheses | 8 |
| 4.3 | Statistical Methods for Effectiveness Analyses | 8 |
| 4.3.1 | Primary Effectiveness Analyses | 8 |
| 5 | Safety Analysis Strategy | 9 |
| 5.1 | Safety Endpoints | |
| 5.2 | Safety Hypotheses | |
| 5.3 | Statistical Methods for Safety Analyses | 10 |
| 5.3.1 | Adverse Events | |
| 5.3.2 | Biomicroscopy Findings/Slit Lamp Examination | |
| 5.3.3 | Device Deficiencies | 11 |

Alcon - Business Use Only Statistical Analysis Plan

Document: TDOC-0055319

Version: 1.0; CURRENT; Most-Recent; Effective

Status: Effective

| 9 | Appendix | 13 |
|-----------|----------------------------------------------|----|
| | List of Tables | |
| Table 1-1 | | 5 |
| Table 0_1 | Schedule of Study Procedures and Assessments | 13 |

Alcon - Business Use Only Statistical Analysis Plan Effective Date: 25-May-2018


Status: Effective

## 1 Study Objectives and Design

## 1.1 Study Objectives

#### PRIMARY OBJECTIVE

The primary objective is to assess

contact lens when worn in an extended wear modality (ie, up to 6 nights of continuous wear) as compared to Biofinity soft contact lens.

## 1.2 Study Description

Key components of the study are summarized in Table 1-1.

Table 1-1 Study Description Summary

| Study Design | Prospective, randomized, controlled, double-masked, contralateral |
|---|---|
| Study Population | Volunteer subjects aged 18 or over who are soft contact lens |
| | wearers, excluding Biofinity habitual wearers, have at least |
| | 3 months of contact lens wearing experience, and who wear their |
| | habitual lenses at least 5 days per week and in an extended wear |
| | modality a minimum of 1 night per week. |
| | . Pregnant |
| | and breastfeeding women are excluded from this study. |
| | Target to complete: 20; Planned to enroll: ~22 |
| Number of Sites | ~2 (US) |
| Test Product | soft contact lenses (LID011121) |
| Control Product | Biofinity® (comfilcon A) soft contact lenses |
| Duration of Treatment | Approximately 6 nights of extended wear |
| Visits | Visit 1, Day 1: Baseline/Dispense |
| | Visit 2, Day 2: 1-Day Follow-Up [24 hours (±4 hours) after Visit 1] |
| | Visit 3, 1 Week: 1-Week Follow-Up/Exit [7 days (-1 day) after |
| | Visit 2] |

#### 1.3 Randomization

A member of the Randomization Programming group at Alcon who is not part of the study team will generate the randomized allocation schedule(s) for study lens assignment.

Version: 1.0; CURRENT; Most-Recent; Effective

Effective Date: 25-May-2018

Status: Effective

Document: TDOC-0055319

Subjects will be randomized in a 1:1 ratio to receive and Biofinity contralaterally in one of the sequences below:

Sequence 1: (OD) / Biofinity (OS) Sequence 2: Biofinity (OD) / (OS)

#### 1.4 Masking

This study is double-masked.



#### 1.5 Interim Analysis

There are no plans to conduct an interim analysis and no criteria by which the study would be terminated early based upon statistical determination.

#### 2 Analysis Sets

### 2.1 Safety Analysis Set

Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. As such, the safety analysis set will include all eyes exposed to any study lenses evaluated in this study. For treatment-emergent safety analyses, eyes will be categorized under the actual study lens exposed at the time of the clinical assessment.

# 3 Subject Characteristics and Study Conduct Summaries

Demographic information (age, sex, ethnicity, and race) and habitual lens information will be tabulated.




Status: Effective



#### 4 Effectiveness Analysis Strategy

This study defines one primary endpoint

Analysis Set will serve as the primary set for all effectiveness analyses.

The Safety

All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation for missing values will be carried out for the primary analysis.

Effective Date: 25-May-2018

## 4.1 Effectiveness Endpoints

#### **Primary Endpoint**

The primary endpoint is distance visual acuity (VA) with study lenses, collected in Snellen, for each eye. Conversion will be made to the logMAR scale.



Version: 1.0; CURRENT; Most-Recent; Effective

Effective Date: 25-May-2018

Status: Effective

### 4.2 Effectiveness Hypotheses

#### **Primary Effectiveness**

Document: TDOC-0055319

No inferences are to be made on the primary effectiveness endpoint; therefore, no hypotheses are formulated.



#### 4.3 Statistical Methods for Effectiveness Analyses

#### 4.3.1 Primary Effectiveness Analyses

Summary statistics will be provided at each visit (Dispense, 1-Day Follow-up, 1-Week Follow-up). Descriptive summary statistics will be displayed with counts and percentages on the Snellen categories, and n, mean, standard deviation, median, minimum, and maximum for the converted logMAR values.



Status: Effective

Version: 1.0; CURRENT; Most-Recent; Effective

Effective Date: 25-May-2018

# 5 Safety Analysis Strategy

Alcon - Business Use Only Statistical Analysis Plan

Document: TDOC-0055319

# 5.1 Safety Endpoints

The safety endpoints are

- Adverse events (AE)
- Biomicroscopy Findings/Slit Lamp Examination
  - Limbal hyperemia
  - Bulbar hyperemia
  - Corneal staining
  - Conjunctival staining
  - Palpebral conjunctival observations
  - Corneal epithelial edema
  - Corneal stromal edema

Effective Date: 25-May-2018 Alcon - Business Use Only Statistical Analysis Plan


Status: Effective

Corneal vascularization

Conjunctival compression/indention

Chemosis

Corneal infiltrates

Other findings

Device deficiencies

#### 5.2 Safety Hypotheses

There are no formal safety hypotheses in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of safety endpoints listed in Section 5.1.

#### 5.3 Statistical Methods for Safety Analyses

The analysis set for all safety analyses is the safety analysis set as defined in Section 2.1. Baseline will be defined as the last measurement prior to exposure to study lenses on Visit 1. Safety variables will be summarized descriptively.

#### 5.3.1 Adverse Events

The applicable definition of an AE is in the study protocol. All AEs occurring from when a subject signs informed consent to when a subject exits the study will be accounted for in the reporting.

Analysis and presentation of pre-treatment AEs will be separated from treatment-emergent AEs occurring during the study period. A pre-treatment AE is an event that occurs after signing informed consent but prior to exposure to the study lens. The period for treatmentemergent AE analysis starts from exposure to study lens until the subject completes or is discontinued from the study.

Descriptive summaries (counts and percentages) for ocular and nonocular AEs will be presented by Medical Dictionary for Regulatory Activities (MedDRA) Preferred Terms (PT). Serious AEs and significant nonserious ocular AEs will be noted. Additionally, relationship to lens will be identified in all AE tables. Unit of presentation for ocular AEs will be eye and nonocular AEs will be subject.

Individual subject listings will be provided for both pre-treatment and treatment-emergent AEs, where any AE leading to study discontinuation will be indicated.

Page 10 Printed By:


Status: Effective

#### 5.3.2 Biomicroscopy Findings/Slit Lamp Examination

Biomicroscopy assessment will be performed at all study visits. The reporting unit for each biomicroscopy finding will be eye.

Effective Date: 25-May-2018

A summary of grade category counts and percentages will be presented for each parameter at each scheduled visit. Findings collected during unscheduled visits will be presented in a subject listing. Furthermore, a listing of "Other" slit lamp findings will also be provided.

#### 5.3.3 Device Deficiencies

A frequency table showing counts for each treatment-emergent Device Deficiency category will be presented. In addition, listings for treatment-emergent and pre-treatment device deficiencies will be provided.



Version: 1.0; CURRENT; Most-Recent; Effective Document: TDOC-0055319 Status: Effective

Effective Date: 25-May-2018

Alcon - Business Use Only Statistical Analysis Plan


Status: Effective



Effective Date: 25-May-2018

# 9 Appendix

Table 9-2 Schedule of Study Procedures and Assessments

| Procedure/ Assessment | Visit 1, Day 1:<br>Baseline/Dispense | Visit 2, Day 2:<br>1-Day Follow-up<br>24 hours after<br>Visit 1 (±4 hours) | Visit 3, Week 1:<br>1-Week<br>Follow-up/Exit<br>7 days (-1 day) of<br>lens wear | Unsched<br>Visit |
|---|---|---|---|---|
| | | | Ideally subjects<br>should be seen<br>within 4 hours of<br>awakening. | |
| Informed Consent | ✓ | - | - | - |
| Demographics | ✓ | - | - | - |
| Medical History | ✓ | - | - | - |
| Concomitant<br>Medications | <b>✓</b> | (✔) | (✓) | (✓) |
| Inclusion/<br>Exclusion | <b>√</b> | - | - | - |
| Habitual lens<br>(brand, power) | ✓ | - | - | - |


Effective Date: 25-May-2018

Status: Effective

| Procedure/ Assessment | Visit 1, Day 1:<br>Baseline/Dispense | Visit 2, Day 2:<br>1-Day Follow-up<br>24 hours after<br>Visit 1 (±4 hours) | Visit 3, Week 1:<br>1-Week<br>Follow-up/Exit<br>7 days (-1 day) of<br>lens wear | Unsched<br>Visit |
|---|---|---|---|---|
| VA w/ habitual<br>correction<br>(OD, OS, Snellen<br>distance)* | <b>√</b> | 1 | <b>√</b> | (✓) |
| | | | <b>↓</b> | |
| Biomicroscopy | <b>√</b> | <b>√</b> ‡ | ✓ at Exit | · · |
| Dispense study lenses | <b>√</b> | - | - | - |
| VA w/ study lenses<br>(OD, OS, Snellen<br>distance) | <b>✓</b> | <b>√</b> | <b>✓</b> | <b>√</b> |
| | | | | • |
| | • | • | _ | _ |
| | | - | I | I |


Status: Effective

| Procedure/ Assessment | Visit 1, Day 1:<br>Baseline/Dispense | Visit 2, Day 2:<br>1-Day Follow-up<br>24 hours after<br>Visit 1 (±4 hours) | Visit 3, Week 1:<br>1-Week<br>Follow-up/Exit<br>7 days (-1 day) of<br>lens wear | Unsched<br>Visit |
|---|---|---|---|---|
| | | - | | |
| | l | | | |
| | ı | | | |
| AEs | ✓ | ✓ | ✓ | ✓ |
| Device deficiencies | ✓ | ✓ | ✓ | ✓ |
| Exit Form | (✓) | (✓) | (✓) | (✓) |

Effective Date: 25-May-2018

<sup>\*</sup>source only

<sup>&#</sup>x27;Comments, optional

<sup>\*</sup>Biomicroscopy with contact lenses still on-eye (not to include corneal staining)

<sup>(✓)</sup> assessment performed as necessary,

Alcon - Business Use Only Statistical Analysis Plan Effective Date: 25-May-2018


Status: Effective